CLINICAL TRIAL: NCT07327320
Title: Comparison of Continuous Norepinephrine and Phenylephrine Infusion for Preventing Hypotension During Low-Dose Spinal Anesthesia in Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Norepinephrine vs. Phenylephrine for Hypotension in Low-Dose Spinal Anesthesia for Cesarean Delivery
Acronym: NORPHE-CD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tam Anh Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TA2.24.03
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Spinal; Cesarean Section; Hypotension, Controlled
Keywords: Norepinephrine; Phenylephrine; Hypotension; Spinal anaesthesia; Cesarean delivery
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: This was a randomized, controlled, single-blind trial with a parallel group design and a 1:1 allocation ratio.
Who Masked: Participant
Masking Description: The randomization sequence was concealed in sequentially numbered, opaque, sealed envelopes. Each envelope contained the specific intervention protocol for the assigned group. The Principal Investigator generated the allocation sequence and prepared the envelopes prior to the study. To ensure concealment, the recruiting investigator opened the next envelope in the sequence only after the participant was enrolled, thereby determining the group assignment.
  This was a single-blind study; only the participants were blinded to the group allocation. Due to the nature of vasopressor administration and the need for real-time hemodynamic management, the investigators and the anesthesiology team were aware of the assigned intervention to ensure patient safety and proper medication delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine (Experimental): Continuous intravenous norepinephrine infusion was administered at 0.05 mcg/kg/min, prepared by diluting 100 mcg in 50 mL of 0.9% sodium chloride
  Interventions: Drug: Norepinephrine
- Phenylephrine (Experimental): Continuous intravenous phenylephrine infusion was administered at 0.25 mcg/kg/min, prepared by diluting 500 mcg in 50 mL of 0.9% sodium chloride
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — Continuous intravenous norepinephrine infusion was administered at 0.05 mcg/kg/min, prepared by diluting 100 mcg in 50 mL of 0.9% sodium chloride
  Arms: Norepinephrine
Drug: Phenylephrine — Continuous intravenous phenylephrine infusion was administered at 0.25 mcg/kg/min, prepared by diluting 500 mcg in 50 mL of 0.9% sodium chloride
  Arms: Phenylephrine

SUMMARY:
This clinical trial was conducted to compare the effectiveness and safety of two medications, norepinephrine and phenylephrine, in preventing hypotension during low-dose spinal anesthesia for cesarean delivery (CD). Although low-dose spinal anesthesia combined with opioids is widely used to mitigate hypotension, the incidence remains unacceptably high. Thus, vasopressors remain essential in maintaining maternal blood pressure during these procedures.

In this study, 100 women were initially assessed, with 2 excluded. The remaining 98 were randomly assigned to receive a continuous infusion of either norepinephrine or phenylephrine. During the follow-up process, 2 patients from each group were lost, resulting in 47 participants per group for final analysis.

The results showed that norepinephrine was significantly more effective, with a lower incidence of hypotension (14.9% vs. 42.6%). It also provided more stable heart rates with fewer episodes of bradycardia and less need for rescue medications. Both treatments were safe for the babies with comparable Apgar scores.

This study suggests that Norepinephrine infusion at 0.05 mcg/kg/min is more effective than phenylephrine at 0.25 mcg/kg/min in preventing hypotension during low-dose SA in CD, providing better hemodynamic stability and fewer episodes of bradycardia

DETAILED DESCRIPTION:
Upon arrival in the operating room, the parturient was monitored using standard American Society of Anesthesiologists monitors, including electrocardiography, pulse oximetry, and invasive arterial BP measurement. A large peripheral vein was cannulated using an 18-gauge intravenous catheter for the administration of fluids and medications. Baseline BP was determined by averaging three measurements taken 2 minutes apart in the supine position before SA. Low-dose SA was performed with 8 mg of bupivacaine (Marcain) combined with 20 mcg of fentanyl and 100 mcg of morphine (Opiphine). At injection, patients received 15 ml/kg of 0.9% saline IV and group-specific vasopressors:

* P group: Continuous intravenous phenylephrine infusion was administered at 0.25 mcg/kg/min, prepared by diluting 500 mcg in 50 mL of 0.9% sodium chloride.
* N group: Continuous intravenous norepinephrine infusion was administered at 0.05 mcg/kg/min, prepared by diluting 100 mcg in 50 mL of 0.9% sodium chloride.

Following SA, patients were placed in a 15° left lateral tilt and administered 4 mg of ondansetron and 4 mg of dexamethasone intravenously. The sensory block was assessed at 10 minutes; a block at or above the xiphoid was considered effective. After placental delivery, uterotonics were administered as prescribed by the obstetrician. Vasopressor infusion was stopped 5 minutes after delivery.

BP and heart rate (HR) were recorded every 2 minutes during the first 30 minutes after SA, then every 5 minutes until the end of surgery. Neonatal HR was monitored continuously, and Apgar scores were assessed at 1 and 5 minutes by a neonatologist.

Management of Hemodynamic Events and Bradycardia Hypotension was defined as systolic blood pressure (SBP) < 90 mmHg or a drop of more than 20% from baseline. Management involved increasing the vasopressor infusion rate by 20%, followed by administration of phenylephrine 50 mcg intravenously if the HR was ≥ 75 bpm, or ephedrine 6 mg IV if HR was < 75 bpm. The infusion rate was returned to baseline once SBP recovered to the target range (80-120% of baseline).

Severe hypotension (SBP < 60% of baseline) was treated using the same approach but with a higher dose of rescue vasopressors: phenylephrine 100 mcg IV or ephedrine 12 mg IV, depending on HR.

In cases of hypertension (SBP > 120% of baseline), the vasopressor infusion was reduced by 50%. If the SBP exceeded 130%, the infusion was temporarily stopped and reinitiated at 50% of the original dose once the SBP returned to the target range.

Bradycardia was defined as a HR of less than 60 bpm. Management of bradycardia was based on the patient's hemodynamic status. If bradycardia occurred without hypotension, the vasopressor infusion was temporarily discontinued, and if the HR recovered to ≥ 60 bpm, the infusion was resumed at 50% of the original dose. Persistent bradycardia (>3 minutes) was treated with atropine 0.5 mg IV, up to 3 doses. If bradycardia was associated with hypotension, ephedrine 6 mg IV was administered.

ELIGIBILITY:
Inclusion Criteria:

* Parturients aged ≥18 years
* Classified as American Society of Anesthesiologists physical status II
* Term singleton pregnancies
* Scheduled for elective CD under SA

Exclusion Criteria:

* Refusal to participate.
* Fetal anomalies or suspected fetal compromise
* Preeclampsia or eclampsia
* Conversion to general anesthesia or use of labor analgesia
* Contraindication to SA
* Preexisting cardiovascular or cerebrovascular disease; chronic hypertension
* Baseline bradycardia
* Current use of cardiovascular or antihypertensive medications
* Body mass index more than 40 kg/m²
* Body weight less than 50 kg or more than 100 kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Hypotension | From the completion of spinal injection until 5 minutes after the neonate is delivered.
  Hypotension was defined as systolic blood pressure (SBP) < 90 mmHg or a drop of more than 20% from baseline.

SECONDARY OUTCOMES:
Bradycardia | From the completion of spinal injection until 5 minutes after the neonate is delivered.
  Bradycardia was defined as a HR of less than 60 beat per minute.
Hypertension | From the completion of spinal injection until 5 minutes after the neonate is delivered
  Hypertension was defined as systolic blood pressure (SBP) > 120% of baseline.
Severe hypotension | From the completion of spinal injection until 5 minutes after the neonate is delivered
  Severe hypotension was defined as systolic blood pressure (SBP) < 60% of baseline
Requirement for rescue vasopressors (phenylephrine or ephedrine) and atropine | From the completion of spinal injection until 5 minutes after the neonate is delivered
  Requirement for rescue vasopressors (phenylephrine or ephedrine) and atropine during vasopressor administration
Nausea and vomiting | From the completion of spinal injection until 5 minutes after the neonate is delivered
  Maternal intraoperative nausea or vomiting during vasopressor administration
Neonatal Apgar Score | At 1 and 5 minutes after birth
  The Apgar score is a standardized clinical assessment tool used to evaluate the physical condition of newborns immediately after birth. The title "Apgar" stands for Appearance, Pulse, Grimace, Activity, and Respiration. In this study, the assessment is performed by a qualified neonatologist. Each of the five criteria is scored from 0 to 2, resulting in a total score ranging from 0 to 10.
  Minimum Value: 0. Maximum Value: 10
  Interpretation:
  Scores 0-3: Critically low; indicates the newborn requires immediate life-saving resuscitation.
  Scores 4-6: Fairly low; indicates the newborn may require some resuscitative measures or close monitoring.
  Scores 7-10: Normal; indicates the newborn is in good to excellent condition. Direction: Higher scores represent a better clinical outcome for the neonate.

CONTACTS AND LOCATIONS:
Locations (1):
- Tam Anh TP. Ho Chi Minh General Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Afolabi BB, Lesi FEA. Regional versus general anaesthesia for caesarean section. Cochrane Database of Systematic Reviews. 2012(10). doi: 10.1002/14651858.CD004350.pub3. PubMed PMID: CD004350. 2. Vallejo MC, Attaallah AF, Elzamzamy OM, Cifarelli DT, Phelps AL, Hobbs GR, et al. An open-label randomized controlled clinical trial for comparison of continuous phenylephrine versus norepinephrine infusion in prevention of spinal hypotension during cesarean delivery. International journal of obstetric anesthesia. 2017;29:18-25. Epub 2016/10/11. doi: 10.1016/j.ijoa.2016.08.005. PubMed PMID: 27720613. 3. Klöhr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta anaesthesiologica Scandinavica. 2010;54(8):909-21. Epub 2010/05/12. doi: 10.1111/j.1399-6576.2010.02239.x. PubMed PMID: 20455872. 4. Herbosa GAB, Tho NN, Gapay AA, Lorsomradee S, Thang CQ. Consensus on the Southeast Asian management of hypotension using vasopressors and adjunct modalities during cesarean section under spinal anesthesia. Journal of Anesthesia, Analgesia and Critical Care. 2022;2(1):56. doi: 10.1186/s44158-022-00084-1. 5. Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, et al. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018;73(1):71-92. Epub 2017/11/02. doi: 10.1111/anae.14080. PubMed PMID: 29090733. 6. Allen TK, George RB, White WD, Muir HA, Habib AS. A double-blind, placebo-controlled trial of four fixed rate infusion regimens of phenylephrine for hemodynamic support during spinal anesthesia for cesarean delivery. Anesthesia and analgesia. 2010;111(5):1221-9. Epub 2010/05/25. doi: 10.1213/ANE.0b013e3181e1db21. PubMed PMID: 20495139. 7. Habib AS. A Review of the Impact of Phenylephrine Administration on Maternal Hemodynamics and Maternal and Neonatal Outc
- See also: Related Info — https://doi.org/10.32895/MPR.25.00043